CLINICAL TRIAL: NCT00858624
Title: Neurophysiology and Pharmacology of Cough Reflex Hypersensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jacky Smith (Other)
Responsible Party: Sponsor-Investigator, Jacky Smith, Reader, University of Manchester
Organization: University of Manchester (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 07/H1004/142
Record Dates: First submitted 2009-03-09; First posted 2009-03-10 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Chronic Cough
Keywords: Cough; Cough reflex; NMDA receptor; central sensitisation
MeSH Terms: conditions — Chronic Cough; Cough | interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Chronic Cough Patients (Active Comparator)
  Interventions: Drug: ketamine
- Healthy Volunteers (Active Comparator)
  Interventions: Drug: ketamine

INTERVENTIONS:
Drug: ketamine — Administration of low dose intravenous ketamine. Dose: 0.075mg/kg over 10 minutes followed by 0.005mg/kg/min over 20 minutes. Given as single infusion.

SUMMARY:
A cough lasting more than 2 months is known as a chronic cough, affecting 12-23% of the adult non-smoking population. Chronic cough has many associated complications including incontinence, muscular chest pains, blackouts and depression. Current treatment is often ineffective in these patients. To develop new medications the investigators need to understand more about the mechanisms that can lead to excessive coughing.

This study plans to compare a group of 12 healthy volunteers and 12 patients with a chronic cough. The investigators hypothesise that that chronic cough patients have a more sensitive cough reflex as a result central nervous system hyper-excitability (central sensitisation). The investigators will measure cough reflex sensitivity before and after administration of ketamine, a medication that blocks an important receptor in the central nervous system.

ELIGIBILITY:
Inclusion Criteria:

Healthy Volunteers:

* Over 18 years old
* Measurable cough reflex sensitivity
* No current or past history of chronic cough or chronic respiratory disease.
* No symptoms of gastro-oesophageal reflux disease, asthma or post-nasal drip.

Chronic Cough Patients

* Over 18 years old
* Chronic persistent cough (> 8 weeks) despite investigation and/or treatment trials for cough variant asthma/post nasal drip and gastro-oesophageal reflux disease.
* Normal CXR
* Normal lung function
* Measurable cough reflex sensitivity

Exclusion Criteria:

* Recent Upper Respiratory Tract Infection (4 weeks)
* Pregnancy/breast feeding
* Current smokers or ex-smokers with < 6 months abstinence or cumulative history of > 10 packyears
* Diabetes Mellitus
* Opiate or ACE Inhibitor use.
* Any centrally acting medication which has the potential to alter cough reflex sensitivity.
* Significant and ongoing chronic respiratory, cardiovascular (in particular hypertension), gastro-intestinal, haematological (porphyria), neurological or psychiatric illness.
* Drug or alcohol abuse
* History of allergy or reaction to ketamine of other NMDA receptor antagonists.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Cough Reflex Sensitivity | 6 months

SECONDARY OUTCOMES:
Upper Oesophageal Pain Thresholds | 6 months
Pain Thresholds Pharynx | 6 months
Pain Thresholds Chest Wall | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- University of Manchester, Education and Research Centre, Wythenshawe Hospital, Manchester, Manchester, United Kingdom